CLINICAL TRIAL: NCT03378440
Title: Psychosocial Predictors of Poor Outcomes After a Knee Arthroplasty: Prospective Observational Study.
Brief Title: Psychosocial Predictors of Poor Outcomes After a Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Barcelona (Other)
Collaborators: Hector Beltran-Alacreu, PhD (Unknown)
Responsible Party: Principal Investigator, Marc Terradas Monllor, Marc Terradas-Monllor, PhD Student, University of Barcelona
Other Study IDs: TKA-02
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore the association between the psychosocial variables: pain catastrophizing, fear of movement, coping skills, pain attitudes, anxiety and depression with postoperative outcomes (pain, health functioning, physical performance, and quality of life) after a knee arthroplasty (KA). The prevalence of KA has increased dramatically during the last two decades, its popularity can be attributed to its evident success regarding pain improvement, deformity correction and disability reduction in knee osteoarthritis subjects. However, only a third of the patients report no functional problems after surgery, the 20% of them are unsatisfied with its functional skills and around a 20% are experiencing pain, high disability degrees and a significant quality of life reduction. This results cannot be fully explained by mechanical processes, surgical procedures or surgery variations, but seems to be related to other psychological aspects. Chronic pain subjects often develop maladaptive thoughts and behaviours (i.e. pain catastrophism, kinesiophobia, activity avoidance) which contribute to make the subject suffer physically as well as emotionally, and affect on the intensity and persistency of pain.

This study is a single centre, prospective observational study of subjects undergoing primary KA. The study is designed and aimed to examine the relationship between postoperative psychosocial factors and the development of post-operative persistent pain and disability.

ELIGIBILITY:
Inclusion criteria:

1. To have sufficient Spanish or Catalan reading, writing and speaking skills to comprehend all explanations and to complete the assessment tools.
2. Be able to provide the informed consent.
3. Be scheduled to undergo in a total or unicompartimental knee arthroplasty.
4. Knee osteoarthritis diagnosis.
5. Patients 18 years old or more.

Exclusion criteria:

1. Patients scheduled to undergo in a total knee arthroplasty because of prostheses replacement, tumor, infection or fracture.
2. Patients scheduled to undergo in a bilateral total knee arthroplasty.
3. Patients that will need another total knee or hip replacement surgery in less than a year regarding the current intervention.
4. Patients with other pathologies with characteristic features of a central sensitization. (i.e. Fibromyalgia)
5. Co-existing other inflammatory or rheumatic conditions (i.e. rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus or ankylosing spondylitis)
6. Co-existing other mental condition and/or major depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Senior subjects with osteoarthritis scheduled for a total knee arthroplasty.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Self-reported Pain | Change from baseline to 1, 3 and 6 months after surgical intervention
  Participants will be asked to rate their pain at resting, walking and flexing their knee on a horizontal 100-mm Visual Analogue Scale (VAS). The horizontal line anchors will be "no pain" and "worst imaginable pain". The VAS is a valid and reliable instrument compared with other pain rating scales, and has been well established in clinical practice and research for measuring pain levels in arthritis populations.
Disability / Limitations | Change from baseline to 1, 3 and 6 months after surgical intervention
  Western Ontario and McMaster University Osteoarthritis Index (WOMAC) (Spanish version) will be used to assess patient´s physical function. This questionnaire can be completed in less than 5 minutes. It's a widely used, reliable, valid and responsive measure of outcome in people with osteoarthritis of the hip or knee.

SECONDARY OUTCOMES:
Self-reported Quality of life | 1 week, 1 month, 3 months and 6 months after surgical intervention
  The spanish version of the Euro Quality of Life 5D-5L (EQ-5D-5L) was used to assess the health related quality of life (HRQL).(10) The EQ-5D-5L consists in two pages: the first one is based on a descriptive system that defines health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories: no problems, slight problems, moderate problems, severe problems, extreme problems.(10) A health state is composed by taking one level for each dimension, and a preference-based scoring function is used to convert the descriptive system to a summary index score (ranging from states worse than dead <0 to full health 1).
Kinesiophobia | 1 week, 1 month, 3 months and 6 months after surgical intervention
  Participants will be asked to complete the Tampa Scale for Kinesiophobia (TSK-11) (Spanish version). TSK-11 is a 11 item self-administered questionnaire used to assess the pain-related fear of movement. The TSK-11 uses a 4-point Likert scale with responses ranging from 1 = totally disagree, to 4 = totally agree. Overall scores range from 11 to 44 indicating a higher degree of pain-related fear of movement when the score is higher.
Pain Attitudes | 1 week, 1 month, 3 months and 6 months after surgical intervention
  Participants will be asked to complete the Spanish version of Survey of Pain Attitudes - Brief (SOPA-B). The SOPA-B is a 30 item self-administered questionnaire which evaluates the pain attitudes and is composed of 7 subscales: solicitude, emotion, medical cure, control, physical harm, disability and medication. This questionnaire uses a 5-point Likert scale with responses ranging from 0 = very false to 4 = very true.
Depression and anxiety | 1 week, 1 month, 3 months and 6 months after surgical intervention
  Participants will be asked to complete the Hospital Anxiety and Depression Scale (HADS) (Spanish version) will be used. The HADS is a 14 item self-administered questionnaire comprised of 2 subscales: depression and anxiety, both composed with 7 items. Each item use a 4-point Likert scale with responses ranging from 0 to 4. Overall scores range from 0 to 21 points for each subscales, and final score is presented using each subscale scores separately. The higher the score, the higher are the anxiety or depression levels.
Range of Motion | 1 week, 1 month, 3 months and 6 months after surgical intervention
  Goniometric assessments of knee will be carried out to assess flexion and extension range of motion.
Pain Catastrophism | 1 week, 1 month, 3 months and 6 months after surgical intervention
  The Spanish version of Pain Catastrophizing Scale (PCS) was used to asses thoughts and feelings related to pain experiences.(9) The PCS is a 13 item self-administered questionnaire composed of 3 subscales: rumination, magnification and helplessness. The PCS uses a 5-point Likert scale with responses ranging from 0 = not at all to 4 = all the time. Overall scores range from 0 to 52 points, the higher the score, the higher is the pain catastrophism level.
Function | 1 week, 1 month, 3 months and 6 months after surgical intervention
  30-Second Chair Stand Test (30sCST) will be use to evaluate patient's functionality on standing, because it is a well-recognized test to detect early declines in functional independence.
Walking Speed | 1 week, 1 month, 3 months and 6 months after surgical intervention
  4 Meters Walking Test (4MWT) will be used to evaluate patient's walking speed.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Maculé-Beneyto, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Iriteb S.L., Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Terradas-Monllor M, Rierola-Fochs S, Merchan-Baeza JA, Pares-Martinez C, Font-Jutgla C, Hernandez-Hermoso JA, Ochandorena-Acha M. Comparison of pain, functional and psychological trajectories between total and unicompartmental knee arthroplasties: secondary analysis of a 6-month prospective observational study. Arch Orthop Trauma Surg. 2024 Dec 12;145(1):32. doi: 10.1007/s00402-024-05710-x. PMID 39666075